CLINICAL TRIAL: NCT00145535
Title: SOLX Titanium Sapphire Laser for Trabeculoplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SOLX, Inc. (Industry)
Responsible Party: Doug Adams, SOLX, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLX41
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2009-07

CONDITIONS: Glaucoma; Glaucoma, Open Angle
Keywords: Glaucoma; Glaucoma, open angle; Intraocular Pressure; Trabeculoplasty; laser; laser, surgery
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Titanium sapphire laser treatment
  Interventions: Device: SOLX Titanium Sapphire Laser (TiSaLT)
- 2 (Active Comparator): Argon laser treatment
  Interventions: Device: Argon Laser Trabeculoplasty (ALT)

INTERVENTIONS:
Device: SOLX Titanium Sapphire Laser (TiSaLT) — Spot laser treatment, ~50 spots over 180°
  Arms: 1
Device: Argon Laser Trabeculoplasty (ALT) — Spot laser treatment, ~50 spots over 180°
  Arms: 2

SUMMARY:
Use of the Titanium Sapphire laser for laser trabeculoplasty to reduce intraocular pressure in patients with poorly controlled intraocular pressure on maximally tolerated medical therapy or prior failed laser trabeculoplasty.

DETAILED DESCRIPTION:
This is a multi-center, outpatient study assessing equivalence of the Titanium Sapphire laser (TiSaLT) to the Argon laser (ALT) in the ability to reduce IOP in patients having primary open angle glaucoma in eyes with poorly controlled IOP on maximally tolerated medications and/or prior failed glaucoma surgery. Approximately 120 patients are to be enrolled in the study, with approximately equal numbers of patients enrolled at each of the investigational sites. The investigational sites are to accrue patients with poorly controlled open-angle glaucoma on maximal tolerated medical therapy and/or patients with previously failed laser trabeculoplasty. One half of the eyes will be randomized to treatment with the Argon laser (ALT) as the concurrent control group and the other half will be treated with Titanium Sapphire (TiSaLT) laser.

ELIGIBILITY:
Inclusion Criteria:Clinical Diagnosis of Open Angle Glaucoma

* Patient is aged 18 years or older, with 2 sighted eyes.
* Eye to be treated have average IOP greater or equal to 22 mmHg, measured at 2 pretreatment visits.
* Eye to be treated either exhibits:
* poorly controlled open angle glaucoma and on maximal tolerated medical therapy
* OR poorly controlled open angle glaucoma and failed previous laser trabeculoplasty (180° available to treat if previous ALT; can treat over previous SLT)

Exclusion Criteria:

Patients are not eligible for enrollment if any of the following exclusion criteria are met:

* Eye to be treated has any of the following:

  1. evidence of glaucoma other than open-angle glaucoma;
  2. severe paracentral or generalized field defect;
  3. any ocular condition that precluded adequate visualization and treatment of the trabecular meshwork.
  4. prior glaucoma surgery other than laser trabeculoplasty or peripheral iridotomy.
* Patient has mental impairment such that he/she could not understand the protocol or is not in a position to provide written informed consent.
* Patient is pregnant.
* Patient might require other ocular surgery within the 6-month follow-up period.
* Patient has a medical history that suggested the potential for complications from TiSaLT.
* Having concurrent treatment with systemic steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2004-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure (IOP) | 1 year

SECONDARY OUTCOMES:
Adverse event frequency | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jan S Peterson, MS, RAC, Study Director — The Emmes Company, LLC
Locations (10):
- United States (5):
  - North Bay Eye Associates, Petaluma, California
  - International Eye Care, Tampa, Florida
  - Glaucoma Associates of New York, New York, New York
  - Texan Eye Care, Austin, Texas
  - Mann Eye Institute, Houston, Texas
- Canada (2):
  - Credit Valley EyeCare, Mississauga, Ontario
  - Institut du Glaucome de Montréal, Montreal, Quebec
- Israel (2):
  - Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
- Hospital Clinico San Carlos de Madrid, Madrid, Spain